CLINICAL TRIAL: NCT04885777
Title: Topical Lidocaine Anesthesia for Nasopharyngeal Sampling: A Double-blind Randomized Placebo-controlled Trial
Brief Title: Topical Lidocaine Anesthesia for Nasopharyngeal Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Abdullah Osman KOCAK, Associate Professor of Emergency Department of Ataturk University, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ataturk University0000
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Nasopharyngeal Sampling; Local Anesthesia
Keywords: Lidocaine; Nasopharyngeal sampling; Coronavirus Disease 2019 Testing
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine group (Active Comparator): One ml of a solution containing 20 mg/ml of lidocaine was applied to each nostril of the participants in the Lidocaine group. Thus, a total of 40 mg of lidocaine, 20 mg for each nostril, was given to the individuals of the Lidocaine group.
  Interventions: Drug: Lidocaine
- Placebo group (Placebo Comparator): The Placebo group received only a total of 2 ml of 0.9% NaCl (one ml for each nostril).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lidocaine — Initially, a nasopharyngeal swab was performed on each group without any intervention. Investigators waited at least one hour for the second sample collection. If the participant was still in pain or felt discomfort due to the first sampling, the waiting time has been extended.
  At the second stage, one ml of a solution containing 20 mg/ml of lidocaine, was applied to each nostril of the participants in the Lidocaine group. Thus, a total of 40 mg of lidocaine, 20 mg for each nostril, was given to the individuals of the Lidocaine group. The second samples were collected after waiting 5 minutes following the administration of the solution.
  Other Names: nasopharyngeal sampling
  Arms: Lidocaine group
Other: Placebo — Initially, a nasopharyngeal swab was performed on placebo group without any intervention. Investigators waited at least one hour for the second sample collection. If the participant was still in pain or felt discomfort due to the first sampling, the waiting time has been extended.
  At the second stage, the Placebo group received only a total of 2 ml of 0.9% NaCl (one ml for each nostril). The second samples were collected after waiting 5 minutes following the administration of the solution.
  Arms: Placebo group

SUMMARY:
Introduction: Nasopharyngeal sampling is widely used in the diagnosis of the Coronavirus Disease 2019 (COVID-19). The aim of this study is to evaluate the effects of topical lidocaine application for nasopharyngeal sampling, on pain perception, the comfort of the patients, and the application difficulty for healthcare staff.

Methods: This study is a prospective randomized placebo-controlled study conducted with 100 healthy volunteers (50 participants in Lidocaine group and 50 participants in Placebo group). Two ml of a solution containing 10 mg/ml of lidocaine was applied to each nostril of the participants in the Lidocaine group, and the same dose of 0.9% NaCl to the Placebo group. Investigators performed two repeated sampling one hour apart. The first sampling was performed before intervention, and the second was performed five-minutes after intervention. Investigators compared the changes in pain intensity and discomfort intensity using two numerical rating scales, the frequency of undesirable reactions, and the judgment of the practitioner staff about the sampling procedure between first and second sampling.

DETAILED DESCRIPTION:
This study is a prospective randomized placebo-controlled study with restricted randomization of an allocation ratio of 1:1. We used Random Allocation Software (RAS) for randomization. The study is conducted following the CONSORT guideline and the tenets of the Declaration of Helsinki we obtained the approval of the Ataturk University Clinical Research Ethics Committee. Also, the written informed consent of all participants will obtained.

ELIGIBILITY:
Inclusion Criteria:

-

The inclusion criteria of the study is:

* being 18 years and older
* volunteering to participate in the study.

Exclusion Criteria:

* The exclusion criteria of the study is:

  * taking analgesic drugs before admission,
  * pregnancy,
  * lactation,
  * having a bleeding disorder, *known allergy to Lidocaine, * previous nasal trauma or operation,
  * having respiratory tract infection symptoms (such as fever, headache, runny nose, sore throat, cough, sneeze, breathlessness),
  * having a chronic disease (diabetes, cancer, heart disease, asthma, COPD, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in the severity of pain during the sampling procedure. | 2 hours
  This outcome will measured via a paper questionnaire that had two Numerical Rating Scale (NRS). The NRSs were 100 mm scales ranging from 0 to 10 (0 as the absence of pain/discomfort and 10 as unbearable pain/discomfort).
Changes in the severity of discomfort during the sampling procedure. | 2 hours
  This outcome will measured via a paper questionnaire that had two Numerical Rating Scale (NRS). The NRSs were 100 mm scales ranging from 0 to 10 (0 as the absence of pain/discomfort and 10 as unbearable pain/discomfort).
Changing the frequency of undesirable reactions | 2 Hours
  Changing the frequency of undesirable reactions during between first and second sample collection. We will record head retraction, holding practitioner staff's hand, grimace, cough, and sneeze as the undesirable reaction during the sampling procedure.
Judgment of the practitioner staff about the sampling procedure | 2 Hours
  We will research the appropriateness and the difficultness of the sample collection procedure, for this outcome. If four steps of the sampling procedure (inserting in the nostril, hitting the back of the nasopharyngeal cavity, rotating five times, and removing) have been completed successfully, it will be defined as the sampling procedure is as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Datas will be sharing via internet.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Carpenter CR, Mudd PA, West CP, Wilber E, Wilber ST. Diagnosing COVID-19 in the Emergency Department: A Scoping Review of Clinical Examinations, Laboratory Tests, Imaging Accuracy, and Biases. Acad Emerg Med. 2020 Aug;27(8):653-670. doi: 10.1111/acem.14048. Epub 2020 Jul 26. PMID 32542934
- [Background] Tolia VM, Chan TC, Castillo EM. Preliminary Results of Initial Testing for Coronavirus (COVID-19) in the Emergency Department. West J Emerg Med. 2020 Mar 27;21(3):503-506. doi: 10.5811/westjem.2020.3.47348. PMID 32223871
- [Background] Petruzzi G, De Virgilio A, Pichi B, Mazzola F, Zocchi J, Mercante G, Spriano G, Pellini R. COVID-19: Nasal and oropharyngeal swab. Head Neck. 2020 Jun;42(6):1303-1304. doi: 10.1002/hed.26212. Epub 2020 Apr 30. PMID 32352180
- [Background] Tsujimoto Y, Terada J, Kimura M, Moriya A, Motohashi A, Izumi S, Kawajiri K, Hakkaku K, Morishita M, Saito S, Takumida H, Watanabe H, Tsukada A, Morita C, Yamaguchi Y, Katsuno T, Kusaba Y, Sakamoto K, Hashimoto M, Suzuki M, Takasaki J, Hojo M, Miyoshi-Akiyama T, Sugiyama H. Diagnostic accuracy of nasopharyngeal swab, nasal swab and saliva swab samples for the detection of SARS-CoV-2 using RT-PCR. Infect Dis (Lond). 2021 Aug;53(8):581-589. doi: 10.1080/23744235.2021.1903550. Epub 2021 Mar 24. PMID 33760699